CLINICAL TRIAL: NCT00168285
Title: Pulmonary Rehabilitation in Interstitial Lung Disease - a Multi-Centre, Single-Blinded Randomised Controlled Trial
Brief Title: Pulmonary Rehabilitation in Interstitial Lung Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Alfred (Other)
Collaborators: La Trobe University (Other); Austin Hospital, Melbourne Australia (Other); Victorian Tuberculosis and Lung Association (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRIDe
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Interstitial Lung Disease
Keywords: Exercise; Pulmonary rehabilitation; Idiopathic pulmonary fibrosis; Connective tissue disorders
MeSH Terms: conditions — Lung Diseases, Interstitial; Motor Activity; Idiopathic Pulmonary Fibrosis; Connective Tissue Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Pulmonary Rehabilitation

SUMMARY:
Interstitial lung disease (ILD) is a highly disabling group of conditions including idiopathic pulmonary fibrosis (IPF), acute and chronic interstitial pneumonias, connective tissue diseases and sarcoidosis. People with ILD frequently experience breathlessness on exertion, which limits their ability to undertake daily activities. People with ILD report very poor quality of life due to low levels of physical functioning and vitality, and high levels of breathlessness and fatigue. There are few treatments for ILD and those that are available have limited impact on quality of life.

The aim of this study is to assess the effects of Pulmonary Rehabilitation, which consists of specialised exercise training for people with lung disease, on exercise capacity and quality of life in people with ILD. We hypothesis that exercise training will result in reduced dyspnoea, improved exercise tolerance and enhanced quality of life.

DETAILED DESCRIPTION:
Interstitial lung disease (ILD) is a highly disabling group of conditions including idiopathic pulmonary fibrosis (IPF), acute and chronic interstitial pneumonias, connective tissue diseases and sarcoidosis. People with ILD frequently experience breathlessness on exertion, which limits their ability to undertake daily activities and reduces health-related quality of life.Available treatments for ILD have proved largely ineffective, offering no improvement in survival and demonstrating only limited impact on quality of life.

Aims of the Research

1. Evaluate the effects of Pulmonary Rehabilitation on exercise capacity and quality of life in patients with ILD
2. Determine the physiological response to Pulmonary Rehabilitation in patients with ILD
3. Determine the relationship between the aetiology and severity of ILD and the effects of Pulmonary Rehabilitation.

Comparisons: 8 weeks exercise training compared to control group (maximal exercise capacity, functional exercise capacity, dyspnoea, quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Ambulant
* Stable medical therapy
* Dyspnoea on exertion following maximal treatment

Exclusion Criteria:

* A history of syncope on exertion
* Too unwell to attend the hospital for exercise training
* Any other comorbidities which would prevent exercise training
* Previous Pulmonary Rehabilitation in the last 12 months

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2005-03; Study Completion 2007-05 (Estimated)

PRIMARY OUTCOMES:
Functional exercise capacity

SECONDARY OUTCOMES:
Maximal exercise capacity
Health-related quality of life
Dyspnoea

CONTACTS AND LOCATIONS:
Overall Officials: Anne E Holland, PhD, Principal Investigator — Alfred Hospital and LaTrobe University; Matthew Conron, MBBS, Principal Investigator — The Alfred; Prue Munro, BAppSc, Principal Investigator — The Alfred; Christine McDonald, MBBS PhD, Principal Investigator — Austin Hospital, Melbourne Australia; Catherine Hill, PhD, Principal Investigator — Austin Hospital, Melbourne Australia
Locations (2):
- Australia (2):
  - Alfred Hospital, Melbourne, Victoria
  - Austin Hospital, Melbourne, Victoria

REFERENCES:
- [Derived] Holland AE, Hill CJ, Conron M, Munro P, McDonald CF. Short term improvement in exercise capacity and symptoms following exercise training in interstitial lung disease. Thorax. 2008 Jun;63(6):549-54. doi: 10.1136/thx.2007.088070. Epub 2008 Feb 1. PMID 18245143